CLINICAL TRIAL: NCT05889715
Title: An Interprofessional-led Model of Care to Prevent and Treat Chronic Diseases Using a Whole Food, Plant-based Nutrition Program in a Primary Care Setting
Brief Title: Assessment of Plant-based Program Using Shared Medical Appointment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Louise L Morrison Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC20220903H
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Disease; Nutrition, Healthy
Keywords: Whole food plant-based nutrition; Primary care setting
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The study will use a single-arm with participants to be enrolled in three groups of 15 each (n=45) into the Green Wellness Program: Plants-2-Plate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Green Wellness Program: Plants-2-Plate (Experimental): The Green Wellness Program:Plants-2-Plate is an established program focusing on whole food plant-based predominant eating pattern in academic primary care setting.The dietary approach includes vegetables, fruits, legumes, whole grains, seeds, nuts in small portion, elimination of all or most of animal foods, and reduction of processed foods. Participants will eat ad libitum. In addition, they will receive support to manage stress, improve quality of sleep, and increase physical activity during the SMA.
  Interventions: Other: Green Wellness Program: Plants-2-Plate

INTERVENTIONS:
Other: Green Wellness Program: Plants-2-Plate — A 6-month, intensive interprofessional program focused on a WFPB predominant eating pattern
  Other Names: Whole food, plant-based program

SUMMARY:
Evaluation of the impact of a whole food, plant-based (WFPB) program using shared medical appointments (SMAs) on reducing cardiovascular risk factors and weight loss in overweight/obese adults with at least one chronic disease

DETAILED DESCRIPTION:
The study will use a single-arm with participants enrolled in three groups of 15 each (n=45) into the Green Wellness Program: Plants-2-Plate, an established program focusing on WFPB predominant eating pattern in an academic primary care setting. The program will offer 14 SMAs in a period of 6 months. Participants will attend the SMA weekly for 3 months, followed by a monthly SMA for the last 3 months of the intervention period. In the first session, participants will receive information about the program, and establish a health goal to be met at the end of the program. Each weekly SMA will have a nutrition education lesson, and feedback from the FNP, RN and RD after a brief assessment on health, medication adjustment, food choices, and shared ideas and experiences among the participants. At the end of the session, participants will set a small health goal to be followed during the week with assistance from the inter-professional team. The WFPB dietary approach includes vegetables, fruits, legumes, whole grains, seeds, nuts in small portion, elimination of all or most of animal foods, and reduction of processed food. Participants will eat ad libitum. In addition, they will receive support to manage stress, improve quality of sleep, and increase physical activity during the SMA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years
* Either overweight (BMI > 25kgm-2) or obese (BMI >30 kgm-2)
* Diagnosis of one or more chronic diseases
* Own a smartphone or tablet that has reliable interned/data access
* Agrees to comply with all study requirements
* Can speak and understand English

Exclusion Criteria:

* Diagnosis of cancer
* Previous participant in Green Wellness program: Plants-2-Plate
* Pregnant or planning to become pregnant
* Breastfeeding
* Concurrent weight loss program
* Plans to leave the city or USA for over 2 weeks within 6 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol from blood chemistry panel | Baseline to 6 months
  Change in Total Cholesterol from program beginning to end
Low Density Lipoprotein (LDL) from blood chemistry panel | Baseline to 6 months
  Change in LDL-cholesterol from program beginning to end
HDL-Cholesterol from blood chemistry panel | Baseline to 6 months
  Change in HDL-cholesterol from program beginning to end
Triglycerides from blood chemistry panel | Baseline to 6 months
  Change in triglycerides from program beginning to end
Tumor necrosis factor-alfa (TNF-α) from blood inflammatory biomarker | Baseline to 6 months
  Change in TNF-α from program beginning to end
Interleukin (IL)-18 measurement from blood test | Baseline to 6 months
  Change in Interleukin (IL)-18 from program beginning to end
C-reactive protein (HsCRP) measurement from blood test | Baseline to 6 months
  Change in HsCRP from program beginning to end
Soluble Intercellular Adhesion Molecule-1 (sICAM1) measurement from blood test | Baseline to 6 months
  Change in sICAM1 from program beginning to end

SECONDARY OUTCOMES:
Adherence to WFPB measurement | Baseline to 6 months
  Pattern of adherence is tracked by a mobile health device by number of days of adherence to program
Physical activity measurement | Baseline to 6 months
  Time spent daily on physical activity daily
Systolic Blood pressure measurement | Baseline to 6 months
  Change in Systolic blood pressure from program beginning to end
Diastolic Blood pressure measurement | Baseline to 6 months
  Change in Diastolic blood pressure from program beginning to end
Waist circumference measurement | Baseline to 6 months
  Change in waist circumference from program beginning to end
Weight measurement | Baseline to 6 months
  Change in weight from program beginning to end

CONTACTS AND LOCATIONS:
Overall Officials: Christiane L Meireles, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- UT Health San Antonio, School of Nursing, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during the trial that underlie the results reported will be shared after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the time of publication with no end date.
Access Criteria: Not yet determined.

REFERENCES:
- [Background] Willett WC, Koplan JP, Nugent R, Dusenbury C, Puska P, Gaziano TA. Prevention of Chronic Disease by Means of Diet and Lifestyle Changes. In: Jamison DT, Breman JG, Measham AR, Alleyne G, Claeson M, Evans DB, Jha P, Mills A, Musgrove P, editors. Disease Control Priorities in Developing Countries. 2nd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2006. Chapter 44. Available from http://www.ncbi.nlm.nih.gov/books/NBK11795/ PMID 21250366
- [Result] US Burden of Disease Collaborators; Mokdad AH, Ballestros K, Echko M, Glenn S, Olsen HE, Mullany E, Lee A, Khan AR, Ahmadi A, Ferrari AJ, Kasaeian A, Werdecker A, Carter A, Zipkin B, Sartorius B, Serdar B, Sykes BL, Troeger C, Fitzmaurice C, Rehm CD, Santomauro D, Kim D, Colombara D, Schwebel DC, Tsoi D, Kolte D, Nsoesie E, Nichols E, Oren E, Charlson FJ, Patton GC, Roth GA, Hosgood HD, Whiteford HA, Kyu H, Erskine HE, Huang H, Martopullo I, Singh JA, Nachega JB, Sanabria JR, Abbas K, Ong K, Tabb K, Krohn KJ, Cornaby L, Degenhardt L, Moses M, Farvid M, Griswold M, Criqui M, Bell M, Nguyen M, Wallin M, Mirarefin M, Qorbani M, Younis M, Fullman N, Liu P, Briant P, Gona P, Havmoller R, Leung R, Kimokoti R, Bazargan-Hejazi S, Hay SI, Yadgir S, Biryukov S, Vollset SE, Alam T, Frank T, Farid T, Miller T, Vos T, Barnighausen T, Gebrehiwot TT, Yano Y, Al-Aly Z, Mehari A, Handal A, Kandel A, Anderson B, Biroscak B, Mozaffarian D, Dorsey ER, Ding EL, Park EK, Wagner G, Hu G, Chen H, Sunshine JE, Khubchandani J, Leasher J, Leung J, Salomon J, Unutzer J, Cahill L, Cooper L, Horino M, Brauer M, Breitborde N, Hotez P, Topor-Madry R, Soneji S, Stranges S, James S, Amrock S, Jayaraman S, Patel T, Akinyemiju T, Skirbekk V, Kinfu Y, Bhutta Z, Jonas JB, Murray CJL. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. JAMA. 2018 Apr 10;319(14):1444-1472. doi: 10.1001/jama.2018.0158. PMID 29634829
- [Result] Campbell EK, Fidahusain M, Campbell Ii TM. Evaluation of an Eight-Week Whole-Food Plant-Based Lifestyle Modification Program. Nutrients. 2019 Sep 3;11(9):2068. doi: 10.3390/nu11092068. PMID 31484341
- [Result] Wright N, Wilson L, Smith M, Duncan B, McHugh P. The BROAD study: A randomised controlled trial using a whole food plant-based diet in the community for obesity, ischaemic heart disease or diabetes. Nutr Diabetes. 2017 Mar 20;7(3):e256. doi: 10.1038/nutd.2017.3. PMID 28319109
- [Result] Yokoyama Y, Levin SM, Barnard ND. Association between plant-based diets and plasma lipids: a systematic review and meta-analysis. Nutr Rev. 2017 Sep 1;75(9):683-698. doi: 10.1093/nutrit/nux030. PMID 28938794
- [Result] Springmann M, Clark MA, Rayner M, Scarborough P, Webb P. The global and regional costs of healthy and sustainable dietary patterns: a modelling study. Lancet Planet Health. 2021 Nov;5(11):e797-e807. doi: 10.1016/S2542-5196(21)00251-5. Epub 2021 Oct 27. PMID 34715058
- [Result] Quek J, Lim G, Lim WH, Ng CH, So WZ, Toh J, Pan XH, Chin YH, Muthiah MD, Chan SP, Foo RSY, Yip J, Neelakantan N, Chong MFF, Loh PH, Chew NWS. The Association of Plant-Based Diet With Cardiovascular Disease and Mortality: A Meta-Analysis and Systematic Review of Prospect Cohort Studies. Front Cardiovasc Med. 2021 Nov 5;8:756810. doi: 10.3389/fcvm.2021.756810. eCollection 2021. PMID 34805312
- [Result] Baden MY, Liu G, Satija A, Li Y, Sun Q, Fung TT, Rimm EB, Willett WC, Hu FB, Bhupathiraju SN. Changes in Plant-Based Diet Quality and Total and Cause-Specific Mortality. Circulation. 2019 Sep 17;140(12):979-991. doi: 10.1161/CIRCULATIONAHA.119.041014. Epub 2019 Aug 12. PMID 31401846
- [Result] Scrafford CG, Bi X, Multani JK, Murphy MM, Schmier JK, Barraj LM. Health Economic Evaluation Modeling Shows Potential Health Care Cost Savings with Increased Conformance with Healthy Dietary Patterns among Adults in the United States. J Acad Nutr Diet. 2019 Apr;119(4):599-616. doi: 10.1016/j.jand.2018.10.002. Epub 2018 Dec 24. PMID 30591404
- [Result] Bolori P, Setaysh L, Rasaei N, Jarrahi F, Yekaninejad MS, Mirzaei K. Adherence to a healthy plant diet may reduce inflammatory factors in obese and overweight women-a cross-sectional study. Diabetes Metab Syndr. 2019 Jul-Aug;13(4):2795-2802. doi: 10.1016/j.dsx.2019.07.019. Epub 2019 Jul 26. PMID 31405709
- [Result] Menzel J, Biemann R, Longree A, Isermann B, Mai K, Schulze MB, Abraham K, Weikert C. Associations of a vegan diet with inflammatory biomarkers. Sci Rep. 2020 Feb 6;10(1):1933. doi: 10.1038/s41598-020-58875-x. PMID 32029816
- [Result] Brathwaite N, Fraser HS, Modeste N, Broome H, King R. Obesity, diabetes, hypertension, and vegetarian status among Seventh-Day Adventists in Barbados: preliminary results. Ethn Dis. 2003 Winter;13(1):34-9. PMID 12723010
- [Result] Kirsh SR, Aron DC, Johnson KD, Santurri LE, Stevenson LD, Jones KR, Jagosh J. A realist review of shared medical appointments: How, for whom, and under what circumstances do they work? BMC Health Serv Res. 2017 Feb 4;17(1):113. doi: 10.1186/s12913-017-2064-z. PMID 28160771
- [Result] Kirsh S, Watts S, Pascuzzi K, O'Day ME, Davidson D, Strauss G, Kern EO, Aron DC. Shared medical appointments based on the chronic care model: a quality improvement project to address the challenges of patients with diabetes with high cardiovascular risk. Qual Saf Health Care. 2007 Oct;16(5):349-53. doi: 10.1136/qshc.2006.019158. PMID 17913775
- [Result] Harland, J., and L. Garton. An update of the evidence relating to plant-based diets and cardiovascular disease, type 2 diabetes and overweight. Nutrition Bulletin. 2016; 41.4 : 323-338.
- [Result] Jaacks LM, Kapoor D, Singh K, Narayan KM, Ali MK, Kadir MM, Mohan V, Tandon N, Prabhakaran D. Vegetarianism and cardiometabolic disease risk factors: Differences between South Asian and US adults. Nutrition. 2016 Sep;32(9):975-84. doi: 10.1016/j.nut.2016.02.011. Epub 2016 Mar 4. PMID 27155957
- See also: Strategic Health Plan of the City of San Antonio — http://www.sanantonio.gov/Portals/0/Files/health/News/Reports/StrategicPlan5-27-2017.pdf?ver=2017-05-30-162509-187